CLINICAL TRIAL: NCT00215553
Title: A Multicenter, Randomized, Controlled Trial Comparing the Safety and Effectiveness of SURFAXIN® (Lucinactant) Delivered Via Bronchopulmonary Segmental Lavage to Standard of Care in Patients With Acute Respiratory Distress Syndrome (ARDS).
Brief Title: KL₄Surfactant Treatment in Patients With ARDS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment and administrative reasons
Sponsor: Windtree Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KL4-ARDS-04
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Results first posted 2012-04-27 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- A.1 Lucinactant (Experimental): 3 30-mL aliquots per bronchopulmonary segment using concentrations of 5, 5, and 10 mg/mL total phopholipids. One re-treatment at 48 hours.
  Interventions: Drug: A.1 Lucinactant
- A.2 Lucinactant (Experimental): 3 30-mL aliquots per bronchopulmonary segment using concentrations of 10, 10, and 10 mg/mL total phospholipids. One lavage re-treatment at 48 hours.
  Interventions: Drug: A.2 Lucinactant
- A.3 Lucinactant (Experimental): 2 50-mL aliquots per bronchopulmonary segment using concentrations of 10 and 20 mg/mL total phospholipids. One lavage re-treatment at 48 hours.
  Interventions: Drug: A.3 Lucinactant
- A.4 Lucinactant (Experimental): 2 50-mL aliquots per bronchopulmonary segment using concentrations of 10 and 20 mg/mL total phospholipids (TPL). One re-treatment at 48 hours. One bolus re-treatment (20 mg/mL TPL) in another 48 hours. A second bolus re-treatment (20 mg/mL TPL) administered 48 hours later.
  Interventions: Drug: A.4 Lucinactant
- B.1 Lucinactant (Experimental): 2 50-mL aliquots per bronchopulmonary segment using concentrations of 10 and 20 mg/mL total phospholipids. One lavage re-treatment at 48 hours.
  Interventions: Drug: B.1 Lucinactant
- B.2 Lucinactant (Experimental): 2 50-mL aliquots per bronchopulmonary segment using concentrations of 10 and 20 mg/mL total phospholipids (TPL). One re-treatment at 48 hours. One bolus re-treatment (20 mg/mL TPL) in another 48 hours. A second bolus re-treatment (20 mg/mL TPL) administered 48 hours later.
  Interventions: Drug: B.2 Lucinactant
- B.3 SoC (Other): Received standard ARDS management and ICU care (Standard of Care [SOC]). Included, but was not limited to, support with oxygen, conventional mechanical ventilation, sedations, and paralysis.
  Interventions: Other: B.3 SoC

INTERVENTIONS:
Drug: A.1 Lucinactant — 3 30 mL aliquots at concentrations of 5, 5, and 10 mg/mL
  Other Names: KL₄Surfactant
  Arms: A.1 Lucinactant
Other: B.3 SoC — Standard ARDS management and ICU care
  Other Names: Negative control
  Arms: B.3 SoC
Drug: A.2 Lucinactant — 3 30 mL aliquots at a concentration of 10 mg/mL each
  Other Names: KL₄Surfactant
  Arms: A.2 Lucinactant
Drug: A.3 Lucinactant — 2 50 mL aliquots at concentrations of 10 and 20 mg/mL
  Other Names: KL₄Surfactant
  Arms: A.3 Lucinactant
Drug: A.4 Lucinactant — 2 50 mL aliquots at concentrations of 10 and 20 mg/mL, with bolus re-treatment allowed
  Other Names: KL₄Surfactant
  Arms: A.4 Lucinactant
Drug: B.1 Lucinactant — 2 50 mL aliquots at concentrations of 10 and 20 mg/mL
  Other Names: KL₄Surfactant
  Arms: B.1 Lucinactant
Drug: B.2 Lucinactant — 2 50 mL aliquots at concentrations of 10 and 20 mg/mL, with bolus re-treatment allowed
  Other Names: KL₄Surfactant
  Arms: B.2 Lucinactant

SUMMARY:
Lung wash with KL₄Surfactant of individual lung segments using a bronchoscope compared to usual care alone consisting primarily of assisted (mechanical) ventilation in patients with acute respiratory distress syndrome(ARDS).

DETAILED DESCRIPTION:
This is a multinational, multicenter, two-part, Phase 2 study that will evaluate the tolerability, safety, and efficacy of KL₄Surfactant in adult ARDS patients when administered by sequential bronchoscopic lavage into each of the 19 bronchopulmonary segments of the lung and as a bolus instillation into each lung.

ELIGIBILITY:
Inclusion Criteria:

* Intubated and required mechanical ventilation support
* Met the criteria for ARDS
* Partial pressure of oxygen/fraction of inspired oxygen (PaO2/FiO2) ≤ 200 mmHg and ≥ 60 mmHg within 60 minutes before randomization
* Mean blood pressure was ≥ 60 mmHg immediately before randomization

Exclusion Criteria:

* Had ARDS due solely to a major trauma
* Was currently participating in another clinical trial or received an experimental drug or device within the previous month
* A woman of childbearing age, unless pregnancy was excluded by a negative urine hCG test or if the subject was surgically incapable of childbearing
* Had a previous episode of ARDS that resolved and then recurred during the current hospitalization
* Had a disease that was sufficiently advanced, in the best judgment of the Principal Investigator, to markedly limit life expectancy to < 6 months
* Was known to have AIDS or symptomatic HIV (CD4 counts <500). Subjects with asymptomatic HIV were not excluded
* Received chemotherapy or radiation within the previous 90 days
* Received an organ transplant other than corneal transplants
* Received, or was currently receiving, immunosuppression therapy within the last 6 months
* Had severe neurological damage or the presence of a disease that was likely to significantly prevent weaning from the ventilator
* Had a best Glasgow Coma Score (GCS) of ≤ 8 or an intracranial pressure ≥ 20 cm H2O prior to the institution of sedatives or paralysis

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2001-05; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Gregory, PhD, Study Director — Windtree Therapeutics
Locations (1):
- Discovery Laboratories, Inc., Warrington, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between May 2001 to February 2006 in hospital ICUs
Groups:
- B.3 SoC: Received standard ARDS management and ICU care. Included, but was not limited to, support with oxygen, conventional mechanical ventilation, sedations, and paralysis.
Period: Overall Study
Arm/Group | A.1 Lucinactant | A.2 Lucinactant | A.3 Lucinactant | A.4 Lucinactant | B.1 Lucinactant | B.2 Lucinactant | B.3 SoC
Started | 5 | 6 | 6 | 5 | 28 | 38 | 36
Completed | 5 | 5 | 4 | 4 | 26 | 32 | 36
Not Completed | 0 | 1 | 2 | 1 | 2 | 6 | 0
Not completed — Adverse Event | 0 | 1 | 2 | 1 | 2 | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A.1 Lucinactant | A.2 Lucinactant | A.3 Lucinactant | A.4 Lucinactant | B.1 Lucinactant | B.2 Lucinactant | B.3 SoC | Total
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 28 | 38 | 36 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Between 18 and 65 years | 2 | 5 | 5 | 5 | 26 | 32 | 32 | 107
  >=65 years | 2 | 1 | 1 | 0 | 2 | 6 | 4 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (24.0) | 50.5 (17.1) | 45.6 (16.0) | 41.6 (6.2) | 46.3 (12.5) | 51.8 (13.0) | 47.3 (12.6) | 48.5 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 4 | 1 | 9 | 22 | 16 | 57
  Male | 2 | 4 | 2 | 4 | 19 | 16 | 20 | 67
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 6 | 5 | 25 | 32 | 23 | 102
  Canada | 0 | 0 | 0 | 0 | 3 | 5 | 9 | 17
  Russian Federation | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Patients Being Alive and Not Receiving Mechanical Ventilation for ≥48 Hours at the End of Day 28.
Time Frame: Through 28 days
Population: In Part A, 5 subjects provided a reasonable cohort to adequately examine the safety of each treatment regimen.
  In Part B, 30 subjects were planned to be enrolled in each treatment group (a total of 90 subjects), enough to calculate the dose response curve.
  Analyses conducted on Intent-to-Treat population (all enrolled subjects).
Measure: Number; unit: participants
Arm/Group | A.1 Lucinactant | A.2 Lucinactant | A.3 Lucinactant | A.4 Lucinactant | B.1 Lucinactant | B.2 Lucinactant | B.3 SoC
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 28 | 38 | 36
participants | 2 | 4 | 4 | 5 | 20 | 26 | 29
Statistical Analysis 1: Comparison: B.1 Lucinactant vs B.2 Lucinactant; Null hypothesis: No difference between treatment groups; Test type: Superiority or Other; p = 0.794, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: B.2 Lucinactant vs B.3 SoC; Null hypothesis: No difference between treatment groups; Test type: Superiority or Other; p = 0.236, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: B.1 Lucinactant vs B.3 SoC; Null hypothesis: No difference between treatment groups; Test type: Superiority or Other; p = 0.396, Cochran-Mantel-Haenszel

2. Secondary Outcome: Mortality
Time Frame: Through 28 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | A.1 Lucinactant | A.2 Lucinactant | A.3 Lucinactant | A.4 Lucinactant | B.1 Lucinactant | B.2 Lucinactant | B.3 SoC
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 28 | 38 | 36
participants | 3 | 2 | 0 | 0 | 4 | 9 | 5
Statistical Analysis 1: Comparison: B.1 Lucinactant vs B.2 Lucinactant; Test type: Superiority or Other; p = 0.346, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: B.2 Lucinactant vs B.3 SoC; Test type: Superiority or Other; p = 0.286, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: B.1 Lucinactant vs B.3 SoC; Test type: Superiority or Other; p = 0.964, Cochran-Mantel-Haenszel

3. Secondary Outcome: Days in ICU
Description: Number of days in ICU
Time Frame: Through 28 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | A.1 Lucinactant | A.2 Lucinactant | A.3 Lucinactant | A.4 Lucinactant | B.1 Lucinactant | B.2 Lucinactant | B.3 SoC
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 28 | 38 | 36
days | 23.4 (7.06) | 20.5 (7.53) | 14.3 (9.81) | 20.0 (2.74) | 15.3 (9.01) | 19.9 (7.66) | 17.4 (8.10)
Statistical Analysis 1: Comparison: B.1 Lucinactant vs B.2 Lucinactant; Test type: Superiority or Other; p = 0.028, ANOVA; ANOVA on ranks
Statistical Analysis 2: Comparison: B.2 Lucinactant vs B.3 SoC; Test type: Superiority or Other; p = 0.147, ANOVA; ANOVA on ranks
Statistical Analysis 3: Comparison: B.1 Lucinactant vs B.3 SoC; Test type: Superiority or Other; p = 0.293, ANOVA; ANOVA on ranks

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | A.1 Lucinactant | A.2 Lucinactant | A.3 Lucinactant | A.4 Lucinactant | B.1 Lucinactant | B.2 Lucinactant | B.3 SoC
Serious Adverse Events (participants affected / at risk) | 4/5 | 2/6 | 1/6 | 0/5 | 10/28 | 19/38 | 13/36
Other Adverse Events (participants affected / at risk) | 5/5 | 6/6 | 6/6 | 5/5 | 24/28 | 37/38 | 31/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A.1 Lucinactant (N=5) | A.2 Lucinactant (N=6) | A.3 Lucinactant (N=6) | A.4 Lucinactant (N=5) | B.1 Lucinactant (N=28) | B.2 Lucinactant (N=38) | B.3 SoC (N=36)
Death NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Multi-organ failure (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Sepsis NOS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anoxic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure NOS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Pneumothorax NOS (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 7 (10) | 0 (0)
Hypotension NOS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke NEC (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Venous thrombosis deep limb (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Necrotising enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia NOS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Empyema NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung abscess NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (exc neonatal) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neurologic examination abnormality (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Agitation aggravated (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxic encephelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polyneuropathy NOS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular arrythmia NOS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gangrene NOS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory gas exchange disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tracheostomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous emphysema (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A.1 Lucinactant (N=5) | A.2 Lucinactant (N=6) | A.3 Lucinactant (N=6) | A.4 Lucinactant (N=5) | B.1 Lucinactant (N=28) | B.2 Lucinactant (N=38) | B.3 SoC (N=36)
Anaemia NOS (Blood and lymphatic system disorders) | 2 | 1 | 2 | 3 | 5 | 8 | 5
Leucocytosis NOS (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1 | 1 | 0 | 0
Thrombocythaemia (Blood and lymphatic system disorders) | 0 (0) | 1 | 0 (0) | 1 | 2 | 3 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 1 | 0 (0) | 0 (0) | 2 | 0 (0)
Bradycardia NOS (Cardiac disorders) | 1 | 1 | 1 | 0 (0) | 2 | 2 | 1
Pulmonary oedema NOS (Cardiac disorders) | 1 | 0 | 0 (0) | 0 (0) | 0 | 1 | 3
Constipation (Gastrointestinal disorders) | 0 (0) | 0 | 1 | 1 | 2 | 1 | 2
Diarrhoea NOS (Gastrointestinal disorders) | 0 (0) | 2 | 2 | 1 | 5 | 4 | 6
Ileus (Gastrointestinal disorders) | 0 (0) | 1 | 0 (0) | 1 | 1 | 2 | 1
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 | 0 (0) | 1 | 0 | 2
Multi-organ failure (General disorders) | 2 | 1 | 0 (0) | 0 (0) | 1 | 2 | 1
Pyrexia (General disorders) | 0 (0) | 1 | 1 | 3 | 3 | 2 | 3
Colitis pseudomembranous (Infections and infestations) | 0 (0) | 0 | 0 (0) | 1 | 1 | 1 | 2
Methicillin-resistant Staphyloccal aureus infection (Infections and infestations) | 1 | 0 (0) | 2 | 0 (0) | 2 | 1 | 1
Pneumonia NOS (Infections and infestations) | 2 | 0 | 0 (0) | 0 (0) | 1 | 3 | 2
Sepsis NOS (Infections and infestations) | 2 | 1 | 0 (0) | 0 (0) | 2 | 4 | 1
Sinusitis NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 3 | 2
Urinary tract infection NOS (Infections and infestations) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 3 | 3
Bacteria NOS sputum identified (Investigations) | 1 | 2 | 0 | 1 | 2 | 0 (0) | 0 (0)
Blood pH decreased (Investigations) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 | 1 | 2
Liver function tests NOS abnormal (Investigations) | 0 (0) | 1 | 1 | 0 (0) | 3 | 2 | 1
Oxygen saturation decreased (Investigations) | 1 | 2 | 3 | 4 | 3 | 5 | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 3 | 2 | 0 (0) | 0 (0) | 0 (0) | 4 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3 | 2 | 1 | 3 | 3 | 4
Confusion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 | 2 | 3
Renal failure NOS (Renal and urinary disorders) | 3 | 1 | 0 (0) | 0 (0) | 4 | 3 | 3
Oliguria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0) | 0 (0) | 0 (0) | 3 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 0 (0) | 7 | 4 | 2
Lung infiltration NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 | 1 | 2 | 6 | 4
Pneumothorax NOS (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 (0) | 1 | 5 | 9 | 5
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 | 0 (0) | 4 | 5 | 2
Dermatitis NOS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 | 1 | 4 | 3 | 5
Pressure sore (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 | 2 | 1 | 1 | 2
Subcutaneous emphysema (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 2 | 2
Tracheostomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 | 0 (0) | 1 | 1 | 2
Hypertension NOS (Vascular disorders) | 0 (0) | 0 (0) | 2 | 1 | 3 | 1 | 4
Hypotension NOS (Vascular disorders) | 0 (0) | 1 | 3 | 1 | 5 | 7 | 5
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days